CLINICAL TRIAL: NCT07165795
Title: Pilot Study to Evaluate the Effect of Transcendental Meditation on Telomere Activity and Well-Being Among Nurse Managers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sarasota Memorial Health Care System (Other)
Collaborators: Florida Atlantic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2288149-1
Record Dates: First submitted 2025-06-30; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Meditation
Keywords: nurse manager; well-being; telomere; meditation
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: This study is a two-group randomized clinical trial (intervention and control groups) pilot study consisting of 30 nurse managers, with 15 nursing managers randomly assigned to each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate TM Instruction (Experimental): This group will receive initial TM instruction within three weeks of baseline assessments with follow-up interventions every 2-4 weeks and an expectation of home practice of two 20min meditation sessions per day.
  Interventions: Behavioral: Transcendental Meditation
- Control Group (delayed instruction) (No Intervention): This group will be eligible to receive TM instruction upon completion of the final 4-month assessments, and asked to continue with routine activities throughout study.

INTERVENTIONS:
Behavioral: Transcendental Meditation — Standard TM instruction by certified TM teachers, including 4 days of initial training (60-90 min/day), then follow-up sessions (60-90 min) every 2-4 weeks.
  Arms: Immediate TM Instruction

SUMMARY:
The objective of this study is to evaluate the impact of a health and coping strategy (Transcendental Meditation, or TM) on Telomere Length and Telomerase Activity (known markers of physiological and psychological stress and aging), Perceived Stress, Work Life Balance, Flourishing, Power as Knowing Participation in Change, and Burnout, among nurse managers.

Aim 1: To evaluate the effects of TM compared to usual care delayed instruction on TL and TA.

Aim 2: To evaluate the effects of TM compared to usual care delayed instruction on work life climate, flourishing, perceived stress, burnout, and power as knowing participation in change.

ELIGIBILITY:
Inclusion Criteria:

* Nurse managers within the Sarasota Memorial Health Care System (SMHCS);
* Stable for at least two months on any prescribed medications (for example, anti-anxiety or anti-depressant medications)

Exclusion Criteria:

* prior instruction in the TM technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Telomere Length | baseline, 1-month, 4-months
  T/S ratio; processed by UCSF Blackburn Labs SOP #104D
Telomerase Activity | baseline, 1-month, 4-months
  (# positive copies/10,000 input cells) ; processed by UCSF Blackburn Labs SOP #104D

SECONDARY OUTCOMES:
Work-Life Climate Scale | baseline, 1-month, 4-months
  (Sexton, et al., 2017); measures work/life balance; responses range from 0-4; survey scores range 0-32, with lower scores reflecting better work/life balance.
Secure Flourishing Index, SFI | baseline, 1-month, 4-months
  (Weziak-Bialowolska et al., 2019); measures multidimensional well-being; survey scores range from 0-120, with higher scores reflecting a higher level of flourishing.
Perceived Stress Scale-10 (PSS10) | baseline, 1-month, 4-months
  (Cohen, 1988); measures the perception of stressful thoughts and feelings in preceding month; responses range from 0-40 with higher scores indicating higher levels of stress.
Maslach Burnout Inventory Human Services Survey for Medical Personnel | baseline, 1-month, 4-months
  (Maslach & Jackson, 1984); Consists of three subscales: Emotional Exhaustion (9-items, score range 0-54, higher scores indicate more emotional exhaustion); Depersonalization (5-items, score range 0-18, higher scores indicate more depersonalization); and Personal Accomplishment (8-items, score range 0-48, higher scores indicate higher level of personal accomplishment).
Power as Knowing Participation in Change (PKPCT) | baseline, 1-month, 4-months
  Barrett (1983, 1984, 2010); Scores range from 48-336 in four subscales with higher scores indicating higher levels of perceived power.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided